CLINICAL TRIAL: NCT02899871
Title: Joint Pain Occurring During Anti-TNF Therapy in Chronic Inflammatory Bowel Disease
Acronym: ArthralgieMICI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2014_843_0016
Record Dates: First submitted 2016-09-05; First posted 2016-09-14 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Inflammatory Bowel Diseases
Keywords: joint pain
MeSH Terms: conditions — Inflammatory Bowel Diseases; Arthralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Control: patients treated with anti-TNF not presenting any joint symptoms.
  Interventions: Other: diagnosis of joint
- case: aetiology of joint symptoms
  Interventions: Other: diagnosis of joint

INTERVENTIONS:
Other: diagnosis of joint — The diagnosis of joint pain will be established by a rheumatologist and completed:
  * If necessary, by a clinically guided radiological assessment (plain x-rays, joint ultrasound, bone and joint MRI).
  * serum assays of the anti-TNF administered, as well as screening for associated antibodies.

SUMMARY:
IBD (inflammatory bowel disease) are associated with various types of joint manifestations, especially inflammatory. Patients with IBD treated with anti-TNF commonly report joint symptoms, with variable expressions and aetiologies, possibly responsible for impaired quality of life, and possibly leading to discontinuation of an effective and validated treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females over the age of 18 years at the time of inclusion
* Patients with IBD (Crohn's disease or ulcerative colitis), diagnosed by a set of compatible clinical (chronic diarrhoea, haematochezia, anoperineal lesions, etc.), laboratory, histological and endoscopic arguments. Patients will be included regardless of the severity of their disease, its clinical course, the type of lesions, and the presence or absence of associated manifestations.
* Patients treated with anti-TNF: infliximab or adalimumab.
* Informed patients not refusing to participate.
* Patients covered by French national health insurance.

Exclusion Criteria:

* Patients under the age of 18 years at the time of inclusion.
* Patients previously treated with anti-TNF, but no longer treated with anti-TNF at the time of inclusion.
* Protected majors (under permanent or temporary guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IBD (Crohn's disease or ulcerative colitis),
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Diagnosis of joint pain | 1 year
  presence or absence : The diagnosis of joint pain will be established by a rheumatologist and completed:
  * If necessary, by a clinically guided radiological assessment (plain x-rays, joint ultrasound, bone and joint MRI).
  * serum assays of the anti-TNF administered, as well as screening for associated antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis DUPAS, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France